CLINICAL TRIAL: NCT05213715
Title: The Effect Of Somatosensory Perception And Proprioception On Upper Extremity Functional Skills In Children With Hemiparetic And Diparetic Cerebral Palsy
Brief Title: The Effect Of Somatosensory Perceptıon And Proprıoceptıon On Upper Extremıty Functıonal Skılls
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSUU
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy; Somatosensory Disorders; Upper Extremity Dysfunction; Proprioceptive Disorders
MeSH Terms: conditions — Cerebral Palsy; Somatosensory Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1/Children with diparetic cerebral palsy: 1/Children with diparetic cerebral palsy
  Interventions: Other: assessment
- 2/Children with hemiparetic cerebral palsy: 2/Children with hemiparetic cerebral palsy
  Interventions: Other: assessment
- 3/healty peer aged children: 3/healty peer aged children
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — assessment of upper extremity functions, somatosensorial functions and proprioseption of upper extremity

SUMMARY:
Cerebral Palsy (CP) is a non-progressive neurodevelopmental disorder characterized by posture and movement disorders as a result of damage to the immature brain for any reason before, during or after birth.In addition to tone, postural and neuromuscular control in children with Cerebral Palsy; Problems are also observed in communication skills, perceptual and cognitive systems and sensory systems.

DETAILED DESCRIPTION:
In neurodevelopmental theory, sensory and motor systems mutually support the development of each other. In addition to the motor problems observed in SP; Sensory-motor impairment, which occurs with the effects of systems such as proprioception, tactile (touch), and vestibular (balance), emerges as the main problem. With the involvement of the central nervous system (CNS) in CP, the sensory systems are also affected along with the motor systems. The involvement of the sensory system is seen in 45% of these children and presents with a white matter lesion. One of the important factors affecting the activities of daily living (ADL) in children with Cerebral Palsy is the deficiencies in their functions as a result of the affected upper extremity. Deficiencies in sensory input can cause delays in learning new motor movements. This can result in disuse of the extremities and sensitivity. The somatosensory cortex, which is important for sensory integration; It is the area of the brain that is sensitive to tactile sensations from the body. It is known that the somatosensory system, which carries these tactile stimuli to the somatosensory cortex, is active from the early stage of life. Sensory and motor interactions experienced in the early stages of life are important for motor development even in the early stages. The improvement in measurable cortical responses of the tactile system; It starts from the 8th week of intrauterine and continues until the postpartum period. In the newborn period, the infant's responses to tactile and proprioceptive stimuli play an important role in the development of motor, cognitive, social and communication skills during infancy and early childhood. The aim of this study is to investigate the effects of somatosensory perception and proprioception on upper extremity functional skills in children with hemiparetic and diparetic CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hemiparetic and Diparetic CP with Gross Motor Function Classification System (GMFCS) Level ≤ 3
* Children with ≤ 2 upper extremity muscles according to the Modified Ashworth Scale (MAS)
* Children with Manual Skills Classification System (MACS) ≤ 3
* Not being diagnosed with mental disability by the RAM (Guidance Research Center)
* Children with CP aged 6-18 years
* Not receiving surgery or Botox (Botulinum Toxin) treatment in the last 6 months
* Children with CP with parental approval

Exclusion Criteria:

* Joint contracture in the shoulder, elbow and hand-wrist
* Having any hearing or vision problems

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children with cerebral palsy and healty peer aged children
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
upper extremity proprioseption test | first day of assessment
  Measurements will be done by a goniometer for bilateral upper extremity shoulder flexion-abduction, elbow flexion-extension, supination-pronation, hand-wrist flexion. The eyes will be closed or the head turned to the opposite direction of the evaluated area. The difference between the value for the full range and the value for the half range will be recorded on the test paper as angular. Higher angular difference indicates worse proprioception.
Kinesthesia Test | first day of assessment
  The difference in the distance between the point where the child ends the movement and the end point of the real line is measured on the evaluation paper with a ruler. The total value of the right and left obtained is recorded by subtracting from 50. The higher the difference, the better the kinesthesia. The test will be applied bilaterally.
somatosensory perception of upper extremity (touch stimulus localization test) | first day of assesment
  Touch stimulus localization test is one of the Ayres' Southern California Sensory Integration and Praxis Test (SIPT) somatosensory perception subtests. Before starting the test, the child is asked to close his eyes. The hand, wrist and forearm are touched once with a pencil in order, first in the pronation position and then in the supination position, and the child is asked to point to the touched area with his finger. The distance between the place touched by the pen and the place indicated by the child is measured with a ruler and recorded on the evaluation sheet in cm. The test is applied bilaterally. Evaluation; The farther the distance between the real touched place and the child touches, the worse tactile perception is interpreted, the closer the real touched place and the child's touched place, the better it is interpreted to show tactile perception.
somatosensory perception of upper extremity (double-touch stimulus localization test) | first day of assesment
  Double-touch stimulus localization test is one of the Ayres' Southern California Sensory Integration and Praxis Test (SIPT) somatosensory perception subtests. Before starting the test, the child is asked to close his eyes. With 2 separate pens, you can simultaneously use two different points such as left hand-right cheek, right hand-left hand, left cheek-right cheek, left hand-left cheek, right hand-left cheek, right hand-right cheek while eyes are closed. tactile. The child is asked to say or show both points touched. If the child knows both points, 2 points, 1 point if he knows one, 0 points if he does not know, and a total score is obtained. In scoring, where the best value is measured out of 14, the lower this value is interpreted as the worse tactile perception, the closer it is to this value, the better tactile perception is interpreted.
somatosensory perception of upper extremity (finger recognition test) | first day of assesment
  Finger recognition test is one of the Ayres' Southern California Sensory Integration and Praxis Test (SIPT) somatosensory perception subtests. Before starting the test, the child is asked to close his eyes. He is asked to put his hands on the table and the child's eyes are closed and 16 different points (8 right hand-8 left hand) are touched with a pencil. They are asked to point to the touched points with their fingers or to express audibly. For each point touched, scoring is done as 1 for a correct answer and 0 for an incorrect answer. The test was performed bilaterally. The patient's total score is obtained by summing the scores for both hands. In this measurement method, which is evaluated out of 16; The closer the value to 16 indicates good tactile perception, while the farther away it is, the worse it indicates tactile perception.
somatosensory perception of upper extremity (right-left discrimination test) | first day of assesment
  Right-left discrimination test is one of the Ayres' Southern California Sensory Integration and Praxis Test (SIPT) somatosensory perception subtests. The child is asked to repeat the same by giving 10 body imitation commands. With the paper with the test questions in the hands of the physiotherapist, the assessment of the child begins. The score for the test is 2 points if he answers correctly in the first three seconds, 1 point if he answers in ten seconds, and 0 points if he fails to answer. The total score is recorded by summing all the sub-scores of the child from the 10 questions in the test.
The Jebsen Taylor Hand Function Test (JTHFT) | first day of assesment
  The Jebsen Taylor Hand Function Test (JTHFT) will be used to assess upper extremity functional skills. JTEFT, which is used in the 6-18 age range, consists of serial subtests representing hand function in daily life. The application of this test, which consists of 6 items, takes 15-45 minutes. A scaled board is used to provide a standard arrangement of objects in the test. The time when all activities are done is recorded with a stopwatch. Higher duration indicates worse hand function.

SECONDARY OUTCOMES:
manuel ability classification system (MACS) | first day of assessment
  It is a classification system created to classify the hand skills of children with CP between the ages of 4-18, such as grasping and releasing objects in daily life, and how they use their hands while holding objects. MACS defines five levels. The higher level indicates worse hand function.
Gross Motor Function Classification System(GMFCS) | first day of assessment
  Gross motor function classification system (GMFCS) is a classification system developed by Palisano et al. in 1997 and expanded in 2007 to classify the gross motor functions of children with CP. Gross motor function in children with CP is a standardized method that classifies motor function differences, especially in sitting and walking, at 5 levels. A higher level indicates worse function.
demographic information | first day of assessment
  demographic information will be recorded (age, gender, height, weight)

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Hatice Adıgüzel, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No